CLINICAL TRIAL: NCT06035718
Title: Comparing the Effectiveness of Transcranial Direct Stimulation (tDCS) and Probiotic Supplementation on Risky Decision-making, Impulsivity, Self-control, and Food Selection in Overweight Adults
Brief Title: Effect of Transcranial Direct Current Stimulation (tDCS) and Probiotic Supplementation in Overweight Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tehran (Other)
Collaborators: University of Messina (Other); Tabriz University (Other)
Responsible Party: Principal Investigator, reza kazemi, Assistant professor, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Overweight
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity
Keywords: transcranial direct current stimulation; obesity; overweight; impulse control
MeSH Terms: conditions — Overweight; Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active tDCS over the dorsolateral prefrontal cortex (DLPFC) (Experimental): In this group, participants will receive active 2 milliampere (mA) tdcs over the DLPFC (anode on F3 and cathode onF4) for 20 minutes.
  Interventions: Device: tDCS
- Active tDCS over the ventromedial prefrontal cortex (VMPFC) (Active Comparator): In this group, participants will receive active 2 mA tdcs over the VMPFC (anode on Fpz and cathode on Cz) for 20 minutes.
  Interventions: Device: tDCS
- Sham tDCS Stimulation (Sham Comparator): In this group, participants will receive sham tDCS which will ramp up for 30 s at the beginning of the session and then ramp down and be switched off during the 20-minute stimulation session.
  Interventions: Device: Sham tDCS
- Probiotic supplementation (Active Comparator): In this group, participants will consume 2 probiotic supplements (The synbiotics family) daily, for one month.
  Interventions: Drug: Probiotic Blend Capsule

INTERVENTIONS:
Drug: Probiotic Blend Capsule — By a probiotic blend capsule a specific product is intended which contains the following: Lactobacillus rhamnosus Lactobacillus plantarum Lactobacillus casei Lactobacillus helveticus Lactobacillus acidophilus Lactobacillus bulgaricus Lactobacillus gasseri Bifidobacterium bifidum Bifidobacterium lactis Bifidobacterium breve Bifidobacterium longum Streptococcus thermophile Fructooligosaccharides (FOS).
  Arms: Probiotic supplementation
Device: tDCS — Using a tDCS device, a mild direct electric current is going to be non-invasively administered to the brain using rubber electrodes placed over the scalp.
  Arms: Active tDCS over the dorsolateral prefrontal cortex (DLPFC); Active tDCS over the ventromedial prefrontal cortex (VMPFC)
Device: Sham tDCS — Using a tDCS device, a mild direct electric current is going to be non-invasively administered to the brain using rubber electrodes placed over the scalp. At this arm the electric current will be applied for a very short time (30 s) after which the device will turn off, thus providing the initial tingling sensation over the scalp but not interfering with the ongoing brain activity.
  Arms: Sham tDCS Stimulation

SUMMARY:
The aim of the current study is to investigate and compare the effectiveness of probiotic supplementation and tDCS stimulation on risky decision-making related to food choices in overweight people. Considering the relatively established communication and interaction between the gut-brain-microbiome axis, the investigators expect that transcranial direct current stimulation and probiotic supplementation can both improve decision-making (decrease risky and impulsive decisions) and increase self-control in overweight people.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 25
* Higher than normal fat level

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Smoking more than 10 cigarettes a day
* Excessive consumption of alcohol
* Suffering from chronic cardiovascular and kidney diseases
* Chronic digestive diseases such as celiac disease,
* Chronic inflammatory bowel diseases such as colitis, intestinal surgery, cancer, etc.
* Suffering from acute and chronic diarrhea in the last one month
* Taking antibiotics in two months before the start of the study,
* Continuous use of prebiotic and probiotic products and drugs in one month before the start of the intervention
* Frequent use of antibiotics during the last month before the start of the intervention
* Taking weight loss medications and following a special slimming diet in the last 3 months before the intervention.
* History of epilepsy and seizures, stroke,
* Use of pacemaker
* Presence of metal implanted in the scalp or brain,
* Presence of skin lesions at the tDCS stimulation site, and history of head injury or brain surgery.
* Brain disorders and long-term and chronic use of neuropsychiatric drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Body analysis test | Depending on the experimental group: 10 stimulation days in tDCS groups and 30 days in the probiotic group.
  This is a technique to determine the percentage of body mass that is fat compared to muscle. It can also indicate where the fat and muscle are carried within the body.
Impulsive Behavior Scale Questionnaire measuring Urgency, Premeditation (lack of), Perseverance (lack of), and Sensation seeking (UPPS) | Depending on the experimental group: 10 stimulation days in tDCS groups and 30 days in the probiotic group.
  This is a self-report tool that assesses five subscales (urgency, premeditation, perseverance, sensation seeking, and positive urgency) that are used to measure five distinct dimensions of impulsive behavior; each scale ranging from 4 to 16); Higher scores represent worse outcome.
Eating attitudes Test (EAT-26) | Depending on the experimental group: 10 stimulation days in tDCS groups and 30 days in the probiotic group.
  This tool is used to identify the presence of "eating disorder risk" based on attitudes, feelings and behaviours related to eating. The total score (between 0 and 78) provides an overall risk score, where higher scores indicating greater risk of an eating disorder.
Balloon analogue risk task (BART) | Depending on the experimental group: 10 stimulation days in tDCS groups and 30 days in the probiotic group.
  BART is a computerized decision-making task that is used to assess risk-taking behavior. The BART simulates a real-world situation, involving actual risky behavior, where taking a risk up until a certain point yields a reward.
Tangney self-control questionnaire (Form 36) | Depending on the experimental group: 10 stimulation days in tDCS groups and 30 days in the probiotic group.
  This is a self-report measurement to assess individual differences in traits of self-control. Scores range from 0 to 144 with higher scores representing worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Heysiattalab, PhD, Study Director — University of Tabriz; Reza Kazemi, PhD, Study Director — University of Tehran; Sara Derafsheh, MSC, Principal Investigator — University of Tabriz
Locations (1):
- Atieh neuroscience center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No